CLINICAL TRIAL: NCT06821685
Title: Clinical Study of Autologous Decidual-like Natural Killer Cells Therapy for Infertility or Adverse Pregnancy History Caused by Abnormal Uterine Natural Killer Cells
Brief Title: Autologous Decidual-like Natural Killer Cells Therapy for Infertility or Adverse Pregnancy History
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: The University of Science and Technology of China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-LCYJ-PY-50
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-06

CONDITIONS: Abortion, Habitual; Infertility Unexplained; Embryo Implantation; Pre-Eclampsia
Keywords: recurrent pregnancy loss; repeated implantation failure; unexplained infertility; decidual natural killer cells
MeSH Terms: conditions — Abortion, Habitual; Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- autologous decidual-like NK cells (Experimental): Autologous decidual like NK cells will be isolated and induced in vitro culture from the patients' peripheral blood and perfused into their uterine.
  Interventions: Biological: autologous decidual-like NK cells

INTERVENTIONS:
Biological: autologous decidual-like NK cells — intrauterine infusion

SUMMARY:
The aim of this study is preliminary exploration of the effectiveness and duration of autologous decidual-like NK cells therapy in improving uterine NK cells dysfunction.

DETAILED DESCRIPTION:
Menstrual blood analysis will be performed on patients with infertility or a history of adverse pregnancy outcomes who have fertility needs. Those with abnormal uterine NK cells function will be screened and given informed consent forms pre-treatment. Collecting peripheral blood from the patients, isolating and inducing in vitro culture to obtain autologous decidual like NK cells which will be perfused into their uterine. Perform continuous menstrual blood analysis within 6 months after the first treatment to assess the improvement of uterine NK cell function. If the function of uterine NK cells improves, enter the stage of attempting pregnancy and follow up pregnancy outcomes; If the function of uterine NK cells does not improve, then autologous decidual like NK cells uterine cavity perfusion therapy will be performed again. NK cells intrauterine infusion will be treated up to 2 times.

ELIGIBILITY:
Inclusion Criteria:

* abnormal uterine NK cell function;
* have one of the following medical history: unexplained recurrent spontaneous abortions (≥2 spontaneous abortions, including biochemical pregnancy), repeated implantation failure (failure of implantation of good-quality embryos in at least two IVF cycles), unexplained infertility, early-onset severe gestational hypertension or early-onset fetal growth restriction;
* have clear fertility desires;
* normal ovarian function or with frozen embryos;
* edometrium thickness measured by vaginal ultrasound before ovulation or at mid-luteal phase >= 7mm;
* 18kg/m^2 < Body mass index < 30kg/m^2;

Exclusion Criteria:

* using progesterone receptor modulator;
* chromosomal karyotype abnormalities in one spouse;
* severe endometriosis, uterine fibroids affecting the shape of the uterine cavity or the size of the whole uterus more than 2 and a half months of pregnancy, uterine malformation, uterine adhesion or thin endometrium;
* uncontrolled autoimmune diseases;
* abnormal blood coagulation function, abnormal liver and kidney function, or other uncontrolled basic diseases (hypertension, diabetes, thyroid disease, etc.) that the researcher access which may affect the progress of the study;
* history of pelvic malignant tumors;
* currently participating in other clinical studies;
* allergic to blood products.

Ages: 22 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Improvement rate of NK cells | 6 months after the first intrauterine infusion therapy
  Improvement rate of NK cells in menstrual blood of patients after intrauterine infusion of autologous decidual like NK cells

SECONDARY OUTCOMES:
Duration of improvement in NK cells | 6 months after the first intrauterine infusion therapy
  Duration of improvement in NK cells in menstrual blood of patients after intrauterine infusion of autologous decidual like NK cells
Clinical pregnancy | 1 year after completion of NK cells therapy
  Ultrasound indicates the presence of a gestational sac and fetal heartbeat in the uterine cavity
Ongoing pregnancy | 1 year after completion of NK cells therapy
  At least 12 weeks of pregnancy, ultrasound indicates that the fetus has cardiac activity and the size of the fetus matches the gestational age
Live birth | 1 year after completion of NK cells therapy
  Delivery of any number of neonates born at 26 or more weeks' gestation with signs of life
preeclampsia | 1 year after completion of NK cells therapy
  The occurrence of preeclampsia during successful ongoing pregnancy after cell therapy
fetal growth restriction | 1 year after completion of NK cells therapy
  The occurrence of fetal growth restriction during successful ongoing pregnancy after cell therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yali Hu, Principal Investigator — The Affiliated Drum Tower Hospital of Nanjing University; Hui Zhu, Principal Investigator — The Affiliated Drum Tower Hospital of Nanjing University
Locations (1):
- The Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China